CLINICAL TRIAL: NCT00135239
Title: Study Care Versus Usual Care for Acute Mechanical Lower Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Dr. Paul Bishop, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: C04-0588
Record Dates: First submitted 2005-08-23; First posted 2005-08-25 (Estimated); Last update posted 2008-06-17 (Estimated); Status verified 2008-06

CONDITIONS: Low Back Pain, Mechanical
Keywords: back; Lower Mechanical Back Pain; Rehabilitation
MeSH Terms: conditions — Low Back Pain

INTERVENTIONS:
Procedure: Study care — All study patients will be assessed initially by a physician in the CNOSP outpatient clinic to confirm that they meet the inclusion/exclusion criteria of the study. Patients receiving the EBC intervention will then receive re-assurance, advice to avoid passive treatments, acetominophen (except where contraindicated) for a period of 2-4 weeks, a four week course of lumbar spine spinal manipulative therapy administered by a CNOSP Chiropractor and advice to return to work in some capacity within eight weeks following the start of treatment. Patients randomized to the UC treatment arm will undergo the treatment(s) recommended by their family physicians.
Procedure: Usual care — Patients randomized to the UC treatment arm will undergo the treatment(s) recommended by their family physicians.

SUMMARY:
The most common work-related injury in British Columbia every year is a lower back injury. The many different treatment options that are available to workers with a back injury have often led to confusion and frustration. New back pain research has shown which combinations of treatments are most helpful, but has also shown that many injured workers in British Columbia do not have these treatments made readily available to them. This research study is designed to accurately determine whether or not providing patients suffering from acute back injuries with a combination of all of these recommended treatments, will improve their function, quality of life and return to work.

DETAILED DESCRIPTION:
Objectives:

To determine if evidence-based care (EBC) is more effective than usual care (UC) in improving the functional status of patients with acute mechanical lower back pain. Our secondary objectives are to determine if EBC is effective in improving patient quality of life or time to return to work.

Research Methodology:

Design: This is a two arm, parallel design, randomized trial. Eligibility: Inclusion criteria are residents of British Columbia with mechanical lower back pain (Quebec Task Force on Spinal Disorders Classification categories 1 or 2) of up to four weeks duration.

Recruitment:

All study patients will be recruited from the patient population currently referred for assessment at the Combined Neurosurgical and Orthopaedic Spine Program (CNOSP) outpatient clinic (OPC).

Randomisation:

Patients will be randomized to receive treatment in either the CNOSP outpatient clinic (EBC) or from their family physicians (UC).

Intervention:

All study patients will be assessed initially by a physician in the CNOSP outpatient clinic to confirm that they meet the inclusion/exclusion criteria of the study. Patients receiving the EBC intervention will then receive re-assurance, advice to avoid passive treatments, acetominophen (except where contraindicated) for a period of 2-4 weeks, a four week course of lumbar spine spinal manipulative therapy administered by a CNOSP Chiropractor and advice to return to work in some capacity within eight weeks following the start of treatment. Patients randomized to the UC treatment arm will undergo the treatment(s) recommended by their family physicians.

Outcomes of Interest:

Primary Outcome: Our primary outcome of interest is the difference in the mean changes in functional improvement at sixteen weeks after the start of treatment, defined as the change in modified Roland Disability (RDQ) scores, between the EBC and the UC patient groups.

Secondary Outcomes: Secondary outcomes of interest are the difference in the mean changes in functional improvement at eight weeks and twenty-four weeks after the start of treatment defined as change in modified Roland Disability (RDQ) scores, differences in time to return to work and differences in the 'Bodily Pain and 'Physical Functioning' domains of the SF-36 questionnaire, between the EBC and the UC patient groups.

Statistical Analysis:

The RDQ scores in the two groups will be compared using the Student's T Test. Analysis of co-variance will be used if necessary to adjust for a difference in baseline functional status using baseline RDQ scores as a co-variate. Time to return to work will be compared using Kaplan Meier survival analysis. A between group comparison of survival will be performed using the log-rank test. SF 36 scores will be normalized and the Bodily Pain" and Physical Functioning scales will be compared between the EBC and UC groups, again using an unpaired t-test and if necessary, analysis of covariance. Estimated sample size: 88 subjects are required based on a two-sided independent T Test. Power + 0.80, alpha + 0.05, mean difference + 3 points, standard deviation + 4.4 and allowing 25% for loss to follow-up.

Non-Scientific Summary:

The most common work-related injury in British Columbia every year is a lower back injury. The many different treatment options that are available to workers with a back injury have often led to confusion and frustration. New back pain research has shown which combinations of treatments are most helpful, but has also shown that many injured workers in British Columbia do not have these treatments made readily available to them. This research study is designed to accurately determine whether or not providing patients suffering from acute back injuries with a combination of all of these recommended treatments, will improve their function, quality of life and return to work.

Relevance:

* Why is this study a high priority for WCB funding?

Lower back injuries remain the single most common category of claim for loss made by injured workers. A recent study has shown that the majority of workers in British Columbia with lower back injuries are now receiving treatments that are inconsistent with internationally developed, evidence-based clinical practice guidelines. In addition, a preliminary research study has shown that many aspects of patient recovery from a lower back injury are enhanced by the use of guideline-recommended treatments when compared with guideline discordant treatments.

The proposed study will accurately determine the value of treating lower back-injured patients with a combination of evidence-based treatments. In addition, the results of this study have the potential to significantly impact many issues that are of key importance to the WCB including improving the quality of life of patients with acute lower back injuries, reducing the use of inappropriate treatments that may promote disability and reducing the costs associated with the treatment of these patients.

* What impact will research outcomes have on BC workplaces?

The outcomes of this research study will help clarify the uncertainty that currently exists with respect to which treatments or combination of treatments, are most helpful for lower back-injured workers. The results of this study have the potential to greatly improve the treatment and/or rehabilitation that these patients are currently receiving in British Columbia, and therefore reduce the disability that is associated with a work-related lower back injury.

ELIGIBILITY:
Inclusion Criteria:

* Residents of British Columbia with mechanical lower back pain
* Acute lower back pain with symptoms lasting 2-4 weeks
* Satisfy the Quebec Task Force Classification of Spinal Disorders Categories 1 and 2

Exclusion Criteria:

* Other significant spinal pathology
* Pregnancy
* Patients with Workers' Compensation Board (WCB) claims
* Persistent pain in other areas of the spine

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2006-01; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
To determine if study-based care (SC) is more effective than usual care (UC) in the treatment of patients with acute mechanical lower back pain after 16 weeks | 16 weeks

SECONDARY OUTCOMES:
To determine if SC is more effective than UC in improving the functional status of patients with acute mechanical lower back pain at 8 weeks and 24 weeks. | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Paul Bishop, MD, Principal Investigator — University of British Columbia
Locations (1):
- Medical Rapid Access Spine Clinic, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] 1. Bigos, S.J.B., O.R.; Braen, G.R.; et al., Clinical practice guideline number 4: Acute low back problems in adults. 1994, Agency for Health Care Policy and Research, Public Service, US Department of Health and Human Services: Rockville, MD. p. 65-0642. 2. Spitzer, W.O., et al., Scientific approach to the assessment and management of activity-related spinal disorders. A monograph for clinicians. Report of the Quebec Task Force on Spinal Disorders. Spine, 1987. 12 (suppl)(7): p. S1-59. 3. Practitioners, R.C.o.G., Clinical guidelines for the management of low back pain. Accessed April 6, 2001. 4. Kendall, N.A., Linton, S.J., Main, C.J., Guide to assessing psychosocial yellow flags in acute low back pain: risk factors for long-term disability and work loss. 1997, Accident Rehabilitation and Compensation Insurance Corporation of New Zealand and the National Health Committee.: Wellington (NZ). 5. Abenhaim, L., et al., The role of activity in the therapeutic management of back pain. Report of the International Paris Task Force on Back Pain. Spine, 2000. 25(4 Suppl): p. 1S-33S. 6. Bogduk, N., Draft evidence based clinical guidelines for the management of acute low back pain. 2000, National Health and Medical Research Council: Australia. 7. (CBO), C.B.v.d.I.T., Consensus Lumbosacrale Radicular Syndrome. June 1995: Utrecht. 8. Ruckenschmerzen, H.-. Empfehlungen zur Therapie von Ruckenschmerzen, Artzneimittelkommission der deutschen Arzteschaft (Treatment guidelines - backache. Drug Committee of German Medical Society). Z Artztl Fortbild Qualitatssich. 1997(91): p. 457-460. 9. Hansen, T.M., Bendix, T., Bunger, C.D., et al., Laenderesmerter Klaringsrapport fra dansk selskap for intern medecin. Ugeskr Laeger, 1996. 158(14 (Suppl)): p. 1-18. 10. Keel, P., Perinin, C.H., Schutz-Petitjean, D., et al., Chronicisation des douleurs du dos: Problematique issues. Rapport final du Programme National de Recherche No. 26B. Bale Editions EULAR. 1996. 11. Manniche, C., ed. Low back pain: Frequency, management and prevention from HTA perspective. 1999, Danish Institute for Health Technology Assessment. 12. Borkan, J., Reis, S., Werner, S. et al., Guidelines for treating low back pain in primary care. 1996, The Israeli Low Back Pain Guideline Group. p. 130: 145-51. 13. Koes, B.W., et al., Clinical guidelines for the management of low back pain in primary care: an international comparison. Spine, 2001. 26(22): p. 2504-13; discussion 2513-4. 14. Hayward, R.S., et al., Canadian physicians' attitudes about and preferences regarding clinical practice guidelines. Cmaj, 1997. 156(12): p. 1715-23. 15. Hayward, R.S., Clinical practice guidelines on trial. Cmaj, 1997. 156(12): p. 1725-7. 16. Basinski, A.S., Evaluation of clinical practice guidelines. Cmaj, 1995. 153(11): p. 1575-81. 17. Steven, I.D. and R.D. Fraser, Clinical practice guidelines. Particular reference to the management of pain in the lumbosacral spine. Spine, 1996. 21(13): p. 1593-6. 18. Burton, A.K. and G. Waddell, Clinical guidelines in the management of low back pain. Baillieres Clin Rheumatol, 1998. 12(1): p. 17-35. 19. Hart, L.G., R.A. Deyo, and D.C. Cherkin, Physician office visits for low back pain. Frequency, clinical evaluation, and treatment patterns from a U.S. national survey. Spine, 1995. 20(1): p. 11-9. 20. Cherkin, D.C., et al., Physician views about treating low back pain. The results of a national survey. Spine, 1995. 20(1): p. 1-9; discussion 9-10. 21. Bishop, P.B. and P.C. Wing, Compliance with clinical practice guidelines in family physicians managing worker's compensation board patients with acute lower back pain. Spine J, 2003. 3(6): p. 442-50. 22. Gonzalez-Urzelai V, P.-E.L., Lopez-de-Munain J, Routine primary care management of acute lower back pain: adherence to guidelines. Eur Spine J, 2003. 12: p. 589-594. 23. Bishop, P., Badii, M., Wing, P., Implementation of clinical practice guidelines in workers compensation board patients with acute mechanical back pain: a prospective randomized trial. Proceedings of the North American Spine Society 17th Annual Meeting. Spine Journal, 2002. 2: p. 62-63S. 24. Bishop, P.W., PC, The Implementation of Clinical Practice Guidelines in Family Physicians Managing Workers' Compensation Board Patients with Acute Lower Back Pain Using Patient Specific Direct Physician to Physician Communication: A Prospective Randomized Trial. Spine, 2003. Submitted. 25. McGuirk, B., et al., Safety, efficacy, and cost effectiveness of evidence-based guidelines for the management of acute low back pain in primary care. Spine, 2001. 26(23): p. 2615-22.